CLINICAL TRIAL: NCT04283838
Title: The Effect of Humanistic Care in Healthcare Workers Participated in the Treatment of Coronavirus Disease 2019
Brief Title: Humanistic Care in Healthcare Workers in Coronavirus Disease 2019
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We cannot enroll enough participants.
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: XJTU2H-WH2
Record Dates: First submitted 2020-02-22; First posted 2020-02-25 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-02

CONDITIONS: Coronavirus Disease 2019
Keywords: coronavirus disease 2019; Humanistic Care; mental health; post-traumatic stress disorder; Healthcare Workers
MeSH Terms: conditions — COVID-19; Psychological Well-Being; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Humanistic care (Experimental): Psychological and physical rehabilitation based humanistic care regimen was used to prevent depression and PTSD in healthcare workers who participated in the treatment of COVID-19.
  Interventions: Behavioral: Humanistic Care

INTERVENTIONS:
Behavioral: Humanistic Care — Psychological and physical rehabilitation based humanistic care regimen

SUMMARY:
As of February 17th, 2020, China has 76396 confirmed cases of coronavirus disease 2019 (COVID-19), including 2348 deaths. The impact factors of clinical outcomes among hospitalized patients still need to be clarified. The healthcare workers faced greater mental and physical pressure under long-term, high-intensity, high-risk working conditions. Investigators aim to evaluate the positive effect of humanistic care for healthcare workers participated in the treatment of COVID-19.

DETAILED DESCRIPTION:
As of February 17th, 2020, China has 76396 confirmed cases of coronavirus disease 2019 (COVID-19), including 2348 deaths. As the national medical team sent to Wuhan, the investigators proposed a psychological and physical rehabilitation based humanistic care regimen generated from experience in treating patients with COVID-19. The healthcare workers faced greater mental and physical pressure under long-term, high-intensity, high-risk working conditions. The investigators want to apply this regimen to the healthcare workers who participated in the treatment of COVID-19, to evaluate the positive effect of humanistic care on preventing depression and post-traumatic stress disorder.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare-personnel who are working for treating COVID-19
* Agree to informed consent

Exclusion Criteria:

* disagree to consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-22 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
Self-rating depression scale | 1 month
  Self-rating depression scale will be finished from healthcare workers by a scale table designed by investigator

SECONDARY OUTCOMES:
Incidence of PTSD | 1 month
  the incidence of post-traumatic stress disorder in healthcare workers

CONTACTS AND LOCATIONS:
Overall Officials: Shouping Gong, MD, PhD, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: No